CLINICAL TRIAL: NCT03884517
Title: An Open, Escalating Phase I Clinical Trial of BAT8003 (for Injection) on the Safety, Tolerability and Pharmacokinetics for Patients With Advanced Epithelial Cancer
Brief Title: Clinical Trial of BAT8003 (for Injection) for Patients With Advanced Epithelial Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Considering that the safety risk will affect the subsequent development, it is decided to terminate the test voluntarily
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BAT-8003-001-CR
Record Dates: First submitted 2019-03-15; First posted 2019-03-21 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Advanced Solid Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- BAT8003 0.2mg/kg (Experimental): BAT8003，0.2mg/kg，intravenous infusion, sample size 1-3
  Interventions: Drug: BAT8003
- BAT8003 0.5mg/kg (Experimental): BAT8003，0.5mg/kg，intravenous infusion, sample size 1-3
  Interventions: Drug: BAT8003
- BAT8003 1mg/kg (Experimental): BAT8003，1mg/kg，intravenous infusion, sample size 3
  Interventions: Drug: BAT8003
- BAT8003 2mg/kg (Experimental): BAT8003，2mg/kg，intravenous infusion, sample size 3
  Interventions: Drug: BAT8003
- BAT8003 4mg/kg (Experimental): BAT8003，4mg/kg，intravenous infusion, sample size 3
  Interventions: Drug: BAT8003
- BAT8003 6mg/kg (Experimental): BAT8003，6mg/kg，intravenous infusion, sample size 3
  Interventions: Drug: BAT8003
- BAT8003 8mg/kg (Experimental): BAT8003，8mg/kg，intravenous infusion, sample size 3
  Interventions: Drug: BAT8003
- BAT8003 10mg/kg (Experimental): BAT8003，10mg/kg，intravenous infusion, sample size 3
  Interventions: Drug: BAT8003
- Amplification group (Experimental): BAT8003，intravenous infusion，choose one proper dose from 0.2、0.5、1、2、4、6、8、10mg/kg
  Interventions: Drug: BAT8003

INTERVENTIONS:
Drug: BAT8003 — Phase 1 dose titration study from BAT8003 0.2mg/kg to 10mg/kg, then choose a proper dose for amplification study based on DLT result

SUMMARY:
The trial is divided into three periods. Dosing will be the first day of each cycle, 21 days per cycle. The first period is the day of first study drug delivery until the 21st day, that is, the first treatment cycle. The DLT observation, exploration of MTD, safety of single administration, tolerance and pharmacokinetics, immunity Original research will happen during this period. The second period is a 2-8 dosing cycle, with multiple doses of tolerance, pharmacokinetics, immunogenicity studies, and preliminary efficacy evaluations. After a 2-4 cycle study, patients with good tolerance and no tumor progression will continue to the 5-8 cycle dosing study. The third period is to expand the study. After exploring the MTD, the investigator and the sponsor can discuss to extend another 10-30 cases in a safe and effective dose group to further study the effectiveness and safety of BAT8003 and its pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or his legal representative signs the informed consent form and fully understands the content, process of the study and possible adverse reactions of the study, and is willing to follow up and image evaluation according to the time specified in the protocol.
2. Age 18-75 years old (including boundary value), gender is not limited;
3. advanced epithelial cancer who are ineffective, unable to receive, or absent from standard treatment, histologically or cytologically confirmed;
4. positive Trop2 expression;
5. At least one measurable tumor lesions according to RECIST 1.1(Evaluation Standard for Solid Tumor Efficacy 1.1);
6. The US Eastern Cooperative Oncology Group (ECOG) scores 0 to 1;
7. Expected survival period ≥ 3 months;
8. proper Laboratory test indicators:
9. Echocardiographic examination of left ventricular ejection fraction (LVEF) ≥ 50%;
10. The treatment for solid cancer has been completed for at least 3 weeks, and has basically recovered from the adverse reactions of previous treatment (≤1 grade according to CTCAE5.0（Common Terminology Criteria for Adverse Events 5.0） standard, except for hair loss);

Exclusion Criteria:

1. Have active hepatitis B (HBV) or hepatitis C (HCV) or syphilis;
2. History of immunodeficiency;
3. Other active infections of clinical significance, based on investigator's judgment;
4. other concurrent, severe, or uncontrollable systemic diseases ;
5. History of moderate or severe dyspnea due to advanced malignancy or its complications or severe pulmonary primary disease, or the need for continuous oxygen therapy, or current interstitial lung disease (ILD) Or pneumonia;
6. clinically significant Cardiovascular abnormalities according to any of the following definitions within 6 months prior to enrollment;
7. The brain or other central nervous system metastasis symptom;;
8. There are ≥ 2 grade peripheral neuropathy according to CTCAE5.0（Common Terminology Criteria for Adverse Events 5.0）;
9. Participated in and received other clinical trials within 4 weeks prior to enrollment;
10. Major surgical treatment within 4 weeks;
11. Used of strong CYP3A4 inhibitors and have not undergone circulatory clearance (less than 3 elimination half-lives) prior to administration of the first clinical study drug;
12. Known allergy to the test drug component, or it is suspected that it may be allergic;
13. Pregnant or lactating women;
14. Alcohol abuse, drug abuse or history of drug abuse in the past 6 months;
15. The investigator believes the patient is not suitable for this trail because of other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
dose-limiting toxicity (DLT) | 3weeks
  safety and tolerability endpoint
maximum tolerated dose (MTD) | 3weeks
  safety and tolerability endpoint
Area under the curve（AUC） | no more than 24weeks
  pharmacokinetic endpoint
Maximum serum drug concentration（Cmax) | no more than 24weeks
  pharmacokinetic endpoint
half-life period（t1/2） | no more than 24weeks
  pharmacokinetic endpoint
Maximum serum drug time（Tmax） | no more than 24weeks
  pharmacokinetic endpoint

CONTACTS AND LOCATIONS:
Overall Officials: jian huang, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China